CLINICAL TRIAL: NCT03212846
Title: Muscle Spasticity Reduction in Children With Cerebral Palsy by Means of Hippotherapy: a Randomized Controlled Trial
Brief Title: Muscle Spasticity Reduction in Children With Cerebral Palsy by Means of Hippotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, David Manuel Lucena Anton, PhD, Clinical Professor, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTS671
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Neuromuscular Diseases in Children; Cerebral Palsy, Spastic; Spasticity, Muscle
Keywords: hippotherapy; cerebral palsy; spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Radomized controlled trial with two groups: intervention group (hippotherapy + conventional treatment) and control group (conventional treatment).
Who Masked: Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Children will receive hippotherapy by a licensed physical therapist. Before riding, stretching and warming exercises of the adductor muscles will be performed. Later, the patient will be seated astride with the therapist behind. In any case, the participant had no control of the horse. Therapist will be responsible for correctly positioning the subject on the horse, but no position changes or active intervention of the subject with the therapist will be made. This positioning consists on achieving the optimal body alignment with neutral pelvis.
  Interventions: Other: Hippotherapy
- Control group (No Intervention): Children will receive the conventional treatment, based on physiotherapy related techniques, such as neurodevelopmental treatment (twice a week).

INTERVENTIONS:
Other: Hippotherapy — Children will receive the hippotherapy treatment, based on horse walking in a regular way led by an experienced leader. Sessions will be performed for 45 minutes once weekly for 12 consecutive weeks in an indoor riding area.
  Arms: Treatment group

SUMMARY:
The aim of this study is to evaluate if a intervention with hippotherapy will improve spasticity for children ages 3-14 who have cerebral palsy. The hip aductors spasticity will be measured using the Modified Ashworth Scale (MAS). The intervention will be performed in addition to traditional treatment.

DETAILED DESCRIPTION:
The main aim of the present study is to determine the effects of hippotherapy on the hip aductors spasticity in children with spastic cerebral palsy. Furthermore, as a secondary objective is to evaluate the changes in Modified Ashworth Scale (MAS) after intervention in children ages 3-14.

ELIGIBILITY:
Inclusion Criteria:

* Primor diagnosis of spastic cerebral palsy
* Children aged 3-14

Exclusion Criteria:

* Children with recent injection of botulinium toxin, surgery, or any planned medical or surgical interventions.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | 12 weeks
  The aim of the scale is to assess muscle tone by the joint range of motion, manually evaluated, and clinically recording passive movements' resistance. Each participant will be examined lying supine on a couch in a relaxed position. The MAS scale is, undoubtedly, the most widely used measure for the quantification of muscular hypertonia. The trunk and the head will be maintained in a neutral position to avoid eliciting tonic neck reflexes, and the passive speed movements will be made in the course of one second. It will be performed in left and right hip, independently, 5 to 8 times to obtain a more reliable result. This modified version adds a 1+ scoring category, in order to register resistance in less than half of the range of motion. Thus, the scores range is from 0 to 4, with 6 choices.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing and Physiotherapy, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No
No provided.

REFERENCES:
- [Background] Casady RL, Nichols-Larsen DS. The effect of hippotherapy on ten children with cerebral palsy. Pediatr Phys Ther. 2004 Fall;16(3):165-72. doi: 10.1097/01.PEP.0000136003.15233.0C. PMID 17057544
- [Background] McGibbon NH, Andrade CK, Widener G, Cintas HL. Effect of an equine-movement therapy program on gait, energy expenditure, and motor function in children with spastic cerebral palsy: a pilot study. Dev Med Child Neurol. 1998 Nov;40(11):754-62. doi: 10.1111/j.1469-8749.1998.tb12344.x. PMID 9881805
- [Background] Whalen CN, Case-Smith J. Therapeutic effects of horseback riding therapy on gross motor function in children with cerebral palsy: a systematic review. Phys Occup Ther Pediatr. 2012 Aug;32(3):229-42. doi: 10.3109/01942638.2011.619251. Epub 2011 Nov 29. PMID 22122355
- [Result] Sterba JA. Does horseback riding therapy or therapist-directed hippotherapy rehabilitate children with cerebral palsy? Dev Med Child Neurol. 2007 Jan;49(1):68-73. doi: 10.1017/s0012162207000175.x. PMID 17209981
- [Result] Zadnikar M, Kastrin A. Effects of hippotherapy and therapeutic horseback riding on postural control or balance in children with cerebral palsy: a meta-analysis. Dev Med Child Neurol. 2011 Aug;53(8):684-91. doi: 10.1111/j.1469-8749.2011.03951.x. Epub 2011 Mar 24. PMID 21729249
- [Result] Kwon JY, Chang HJ, Lee JY, Ha Y, Lee PK, Kim YH. Effects of hippotherapy on gait parameters in children with bilateral spastic cerebral palsy. Arch Phys Med Rehabil. 2011 May;92(5):774-9. doi: 10.1016/j.apmr.2010.11.031. PMID 21530725
- [Result] McGibbon NH, Benda W, Duncan BR, Silkwood-Sherer D. Immediate and long-term effects of hippotherapy on symmetry of adductor muscle activity and functional ability in children with spastic cerebral palsy. Arch Phys Med Rehabil. 2009 Jun;90(6):966-74. doi: 10.1016/j.apmr.2009.01.011. PMID 19480872